CLINICAL TRIAL: NCT05880030
Title: The Effect of Supplementation of Vitamin D3 on Inflammation Induced by 100 km Running, Iron Metabolism and Erythropoiesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AWFiS/2022_2_MK
Record Dates: First submitted 2022-12-15; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-11

CONDITIONS: Inflammation; Muscle; Iron Metabolism; Ineffective Erythropoiesis; Healthy
Keywords: Vitamin D; Running; inflammations; erythropoietin; iron; hepcidin
MeSH Terms: conditions — Myositis, Inclusion Body; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Both groups took drops from the same dark bottles, 20 drops per day for two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D (Active Comparator): Vigantol 10 000 IU/day (20 droplets) two weeks supplementation (vitamin D3)
  Interventions: Drug: Cholecalciferol
- Control (Placebo Comparator): sunflower oil, (20 droplets) two weeks supplementation.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Cholecalciferol — cholecalciferol 10000 UI
  Other Names: Vitamin D3
  Arms: Vitamin D
Other: placebo — sunflower oil
  Arms: Control

SUMMARY:
A group of runners received vitamin D (10,000 IU - international unit per day) for two weeks. The aim of the intervention was to check the effect of vitamin D supplementation on selected parameters of inflammation and iron metabolism in comparison with the placebo group. Blood was collected before and after supplementation. Next: before, after 25, 50, 75,100 km running and 12 hours after the run. The data were subjected to statistical analysis.

DETAILED DESCRIPTION:
Subjects were randomized to two groups: the experimental one, n = 20 and the placebo one, n = 20 with the same age, experience in running and 25(OH)D level. The experimental group received vitamin D3 supplementation (around 10,000 UI/day, i.e., 20 droplets -Vigantol medicament, Merck) and the control group received a placebo (20 droplets of sunflower oil, placed in an identical bottle as vitamin D3) for two weeks before a run. The last vitamin D dose was taken 24 h before the 100 km ultra-marathon. 40 male athletes took part in the 100 km ultra-marathon. Blood was collected before (day 0) and after supplementation (day 14). Next (day 15): before, after 25, 50, 75,100 km running and 12 hours after the run (day 16). The data were subjected to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* male
* athletes running ultra-marathons

Exclusion Criteria:

* vitamin D3 supplementation
* multivitamin and iron supplementation
* serum 25(OH)D low < 10 ng/mL
* serum 25(OH)D high > 100 ng/mL
* haemoglobin < 10 g/dL
* other (sports injury, tournament)

Ages: 28 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The change in vitamin 25(OH)D level after two-week supplementation. | Day 0 to day 14
  Measured parameter: vitamin 25(OH)D [ng/ml].
The change in parathyroid hormone level after two-week supplementation. | Day 0 to day 14
  Measured parameter: parathyroid hormone [pg/ml].
Observation of changes in inflammatory parameters:interleukin-6 induced by a 100 km run | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameter of inflammatory: interleukin-6 [pg/ml]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in inflammatory parameters: C reactive protein - CRP induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameter of inflammatory: CRP[mg/l]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in creatine kinase level induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameter: creatine kinase [U/l]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in leucocytes induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameters of inflammatory: leukocytes [G/l]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).

SECONDARY OUTCOMES:
Observation of changes in hepcidin level induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameters of iron metabolism: hepcidin [ng/mL]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in serum iron level induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured serum iron level [µg/dL].Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in ferritin induced by 100 km running. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured parameters of iron metabolism: ferritin [ng/mL]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12h after the run (06 11 2016).
Observation of changes in erythrocytes level induced by a 100 km run. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured erythrocytes level [T/l].Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12 hours after the run (06 11 2016).
Observation of changes in reticulocytes induced by a 100 km run. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured reticulocytes [promil]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12 hours after the run (06 11 2016).
Observation of changes in hematocrit induced by a 100 km run. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured hematocrit [%].Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12 hours after the run (06 11 2016).
Observation of changes in erythropoietin level induced by a 100 km run. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured erythropoietin level [mIU - milli-International unit/mL]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12 hours after the run (06 11 2016).
Observation of changes in erythroferrone level induced by a 100 km run. | Day "15 - the run" and day "16 - 12 hours after the run"
  Measured erythroferrone level [pg/ml]. Collected blood samples before and after 25, 50, 75 and 100-km run (05 11 2016) and 12 hours after the run (06 11 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Kasprowicz, PhD, Study Chair — Gdansk University of Physical Education and Sport

IPD SHARING:
Plan to Share IPD: No